CLINICAL TRIAL: NCT04158973
Title: Bleeding Risk Guided VTE Prophylaxis Strategy for Hospitalized Patients With Lung Cancer: Rationale and Design for a Multicenter, Adjudicator-blinded, Parallel, Randomized Clinical Trial in China
Brief Title: CHIPs-VTE Study in Hospitalized Patients With Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhenguo Zhai,MD,PhD, Principal investigator, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHIPs-VTE in lung cancer
Record Dates: First submitted 2019-09-04; First posted 2019-11-12 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-08

CONDITIONS: Venous Thromboembolic Disease; Pulmonary Embolism; Deep Venous Thrombosis
MeSH Terms: conditions — Pulmonary Embolism; Venous Thrombosis | interventions — Hospitals

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VTE prophylaxis based on bleeding risk assessment (Experimental): Patients will undergo a bleeding risk assessment to determine their entering VTE prophylaxis. Low bleeding risk patients will have once daily sc LMWH prophylaxis. Intermediate bleeding risk patients will have q 12 h sc low dose unfractionated heparin prophylaxis. High bleeding risk patients will have mechanical prophylaxis. Assigned prophylaxis can be interrupted as clinical judgement requires, e.g., for peri-procedural reasons. When patients are discharged, if they have low risk of bleeding at the time of discharge, whatever their bleeding risk assessment at the time of randomization, will begin 5 mg rivaroxaban prophylaxis (two 2.5 mg tablets) once daily with food, starting on the day of discharge, for 15 days.
  Interventions: Other: Bleeding-risk based prophylaxis strategy during hospitalization and extended pharmacological treatment after discharge
- Routine VTE prophylaxis in local clinical practice (Active Comparator): VTE risk assessment and prophylaxis if indicated during hospitalization according to current policies for hospitals in China but no further treatment prophylaxis after discharge.
  Interventions: Other: Routine VTE prophylaxis in hospital

INTERVENTIONS:
Other: Bleeding-risk based prophylaxis strategy during hospitalization and extended pharmacological treatment after discharge — At admission, patents undergo bleeding risk assessment and receive prophylaxis according to bleeding risk. After discharge, they will undergo an extended treatment of 5mg Rivaroxaban once daily for 15 consecutive days,
  Arms: VTE prophylaxis based on bleeding risk assessment
Other: Routine VTE prophylaxis in hospital — Patients randomized to the standard treatment (Control) group will receive routine VTE prophylaxis according to current guidelines and clinical practices, VTE risk assessment and prophylaxis if indicated during hospitalization according to current policies for hospitals in China but no further treatment prophylaxis after discharge
  Arms: Routine VTE prophylaxis in local clinical practice

SUMMARY:
Venous thromboembolism (VTE) is a common complication of malignancies, in particular to lung cancer. Patients with lung cancer in surgical and medical departments are at high risk of VTE development. Prophylaxis is one major way to to prevent it. Currently, VTE prophylaxis is mainly based on VTE-risk assessment. However, all patients hospitalized for cancer are at intermediate or high risk of VTE but their bleeding risk vary. To improve effect of VTE prophylaxis and reduce bleeding events in patients with lung cancer, we will conduct an open-label parallel randomized clinical tria to assess the effect of bleeding risk based prophylaxis strategy among lung cancer patients. We hypothesize that VTE prophylaxis based on bleeding risk assessment with a short post-discharge treatment course is superior to VTE propohylaxis based on VTE risk assessment among hospitalized patients with lung cancer

A sample of 3200 eligible patients will be randomized into experimental or control group with an allocation rate of 1:1. Stratified by medical/surgical units, block randomization with a varying block size of 4 or 6 will be adopted to randomize patients into experimental or control group. In experimental group, patients will undergo bleeding risk assessment and receive prophylaxis according to bleeding risk during hospitalization, and they will also receive an extended pharmacological prophylaxis of 5mg Rivaroxaban once daily for up to 15 consecutive days after discharge. In control group, patients will receive routine VTE prophylaxis, VTE risk assessment and prophylaxis if indicated during hospitalization according to current policies for hospitals in China but no further treatment prophylaxis after discharge.

Patients in both groups will be followed up for 30 days. The primary outcome is symptomatic and asymptomatic objectively proven VTE (deep vein thrombosis (DVT) and/or pulmonary embolism (PE)) within 30 days after initiation of randomization. Ultrasound and CTPA will be performed to detect DVT and PE, respectively. Clinically relevant bleeding (non-major clinically relevant and major bleeding, HIT) and death are secondary outcomes.

DETAILED DESCRIPTION:
Randomization and sequence generation A computerized random-number generator will be used to generate the allocation sequence. In this multicenter trial involving 10 hospitals, randomization procedures will be organized centrally.

Stratified block randomization with a varying block size of 4 or 6 will be used to allocate patients into experimental or control group. Patients with lung cancer will be stratified into those under planned medical or surgical treatments.

In each stratum, patients will be blocked according to their admission sequence. Four or six patients consecutively admitted will be one block depending on the block size. In each block, patients will be randomly allocated into experimental or control group according to sequence generated in advance by software.

Allocation concealment/Blinded randomization Patient assignments will be enclosed in a sequentially numbered, opaque, sealed envelopes (SNOSE). Clinicians in charge of patient enrollment will not know the allocation sequence until eligible patients who meet inclusion and exclusion criteria are enrolled.

An independent statistician will generate the random allocation sequence. Physicians will enroll participants and assign interventions in experimental or control group.

Blinding/Open label This is an open-label trial that patients, clinicians and researchers will know allocation assignments after enrollment. But imaging experts providing the duplex ultrasound and CTPA results will be blinded in order to objectively assess the 30-day CTPA-proven VTE incidence and other outcomes in both groups. An independent data monitoring board will evaluate the trial data and safety.

ELIGIBILITY:
Patients with primary lung cancer admitted to medical units (for chemotherapy, complications, etc) or to surgical units for operations.

Inclusion criteria

1. Aged ≥40 years
2. Have an expected hospital stay ≥72 hours for medical and/or surgical treatment
3. Confirmed lung cancer at admission or proven lung cancer within prior 6 months
4. Evidence of active lung cancer within 6 prior months
5. Written informed consent

Exclusion criteria Patient-related criteria

1. Pregnancy or breastfeeding
2. Inability to be followed-up at until 3 months after randomization
3. have participated in similar trials or are undergoing other clinical trials
4. refuse or are unable to give informed consent VTE/bleeding-related criteria
5. Incidental VTE identified on spiral CT scans which are ordered primarily for staging the malignancy at or any time before enrollment
6. Neurosurgery, vascular procedures, orthopedic surgery intended during the admission
7. Severe renal failure not receiving dialysis (creatinine clearance [CrCl] <30 mL/min), moderate to severe liver dysfunction, severe anemia
8. Uncontrolled hypertension (systolic blood pressure [BP] >180 mmHg, diastolic BP >110 mmHg)
9. severe platelet dysfunction or inherited bleeding disorder (such as haemophilia and von Willebrand's disease)
10. Acute stroke or recent stroke (within 4 weeks)
11. Recent major bleeding (within 3 months)
12. Requiring a full dose of anticoagulant treatment (e.g., recent VTE, atrial fibrillation)
13. Contraindication to heparin or rivaroxaban, e.g., heparin induced thrombocytopenia or history of documented episode of heparin or LMWH induced thrombocytopenia and/or thrombosis (HIT, HAT, or HITTS); recent central nervous system (CNS) bleed, hemorrhagic CNS metastases; active major bleeding with more than 2 units transfused in 24 hours.
14. Contraindication to mechanical prophylaxis, e.g., acute deep vein thrombosis, severe arterial insufficiency (pertains to graduated compression stockings only)
15. Concurrent use of anticoagulants known to increase the risk of bleeding (such as warfarin with INR>2).

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3200 (Estimated)
Dates: Start 2021-12-01 (Estimated); Primary Completion 2022-04-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of symptomatic and asymptomatic objectively proven VTE | 30 days after randomization
  PE incidence detected by CTPA and/or DVT by ultrasound

SECONDARY OUTCOMES:
All-cause mortality | 30 days after randomization
  All-cause deaths that occur during study
Clinically relevant bleeding | 30 days after randomization
  Bleeding that occur in the study
Adverse events | 30 days after randomization
  Safety events related to drug use

CONTACTS AND LOCATIONS:
Overall Officials: Zhenguo Zhai, Doctor, Principal Investigator — China-Japan Friendship Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vitale C, D'Amato M, Calabro P, Stanziola AA, Mormile M, Molino A. Venous thromboembolism and lung cancer: a review. Multidiscip Respir Med. 2015 Sep 15;10(1):28. doi: 10.1186/s40248-015-0021-4. eCollection 2015. PMID 26380084
- [Background] Connolly GC, Dalal M, Lin J, Khorana AA. Incidence and predictors of venous thromboembolism (VTE) among ambulatory patients with lung cancer. Lung Cancer. 2012 Dec;78(3):253-8. doi: 10.1016/j.lungcan.2012.09.007. Epub 2012 Sep 29. PMID 23026639
- [Background] Zhang Y, Yang Y, Chen W, Guo L, Liang L, Zhai Z, Wang C; China Venous Thromboembolism (VTE) Study Group. Prevalence and associations of VTE in patients with newly diagnosed lung cancer. Chest. 2014 Sep;146(3):650-658. doi: 10.1378/chest.13-2379. PMID 24676401
- [Background] Song C, Shargall Y, Li H, Tian B, Chen S, Miao J, Fu Y, You B, Hu B. Prevalence of venous thromboembolism after lung surgery in China: a single-centre, prospective cohort study involving patients undergoing lung resections without perioperative venous thromboembolism prophylaxisdagger. Eur J Cardiothorac Surg. 2019 Mar 1;55(3):455-460. doi: 10.1093/ejcts/ezy323. PMID 30289479
- [Background] Lyman GH, Kuderer NM; American Society of Clinical Oncology. Prevention and treatment of venous thromboembolism among patients with cancer: the American Society of Clinical Oncology Guidelines. Thromb Res. 2010 Apr;125 Suppl 2:S120-7. doi: 10.1016/S0049-3848(10)70029-3. No abstract available. PMID 20433991
- [Background] Zhai Z, Kan Q, Li W, Qin X, Qu J, Shi Y, Xu R, Xu Y, Zhang Z, Wang C; DissolVE-2 investigators. VTE Risk Profiles and Prophylaxis in Medical and Surgical Inpatients: The Identification of Chinese Hospitalized Patients' Risk Profile for Venous Thromboembolism (DissolVE-2)-A Cross-sectional Study. Chest. 2019 Jan;155(1):114-122. doi: 10.1016/j.chest.2018.09.020. Epub 2018 Oct 6. PMID 30300652